CLINICAL TRIAL: NCT06742983
Title: Healing Efficacy of Isobutyl Cyanoacrylate High Viscous Solution in Treatment of Traumatic Ulcer in Children: A Clinical and Experimental Study
Brief Title: Healing Efficacy of Isobutyl Cyanoacrylate High Viscous Solution in Treatment of Traumatic Ulcer in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 402/2021
Record Dates: First submitted 2024-12-15; First posted 2024-12-19 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2024-09

CONDITIONS: Ulcer
Keywords: ulcer; chlorhexidine; Isobutyl cyanoacrylate
MeSH Terms: conditions — Ulcer | interventions — Bucrylate; Chlorhexidine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Isobutyl cyanoacrylate (Experimental): Thin layers of a high viscosity isobutyl cyanoacrylate high viscous solution (periacryl 90 H.V) tissue adhesive will be applied on the ulcer site by using a pipette then rinsed with saline by using another pipette at least three times with an interval of at least 30 seconds once during the treatment episode to allow for complete polymerization, until achieving hemostasis
  Interventions: Other: Isobutyl cyanoacrylate
- Chlorhexidine 0.2% (Experimental): Application of chlorhexidine 0.2% (Elugel 2%) on finger tip then spread it on the ulcer site and gentle massaging twice daily for 9 days
  Interventions: Other: Chlorhexidine (0.2%)
- normal saline (Placebo Comparator): will be treated with cotton soaked with normal saline on the ulcer site 5 times per day
  Interventions: Other: Normal Saline (0.9% NaCl)

INTERVENTIONS:
Other: Isobutyl cyanoacrylate — Thin layers of a high viscosity isobutyl cyanoacrylate high viscous solution Thin layers of a high viscosity isobutyl cyanoacrylate high viscous solution
  Other Names: periacryl 90 H.V
  Arms: Isobutyl cyanoacrylate
Other: Chlorhexidine (0.2%) — Chlorhexidine Digluconate 0.2%
  Other Names: Elugel 2%
  Arms: Chlorhexidine 0.2%
Other: Normal Saline (0.9% NaCl) — Sodium chloride 0.9%
  Other Names: Saline
  Arms: normal saline

SUMMARY:
30 children with traumatic oral ulcer that will be divided into equal three groups. Group A (Isobutyl cyanoacrylate) includes children will be treated with isobutyl cyanoacrylate high viscous solution only once during the treatment episode, group B (control positive) includes children will be treated chlorohexidine gel (0.2%) twice daily and group C (control negative) includes children will be treated with normal saline five times per day. Clinical follow up will be done by assessment of pain perception, photographs of the ulcer will be recorded by using digital camera and measurement of ulcer size in the 1st ,5th and 9th days after treatment

DETAILED DESCRIPTION:
Thirty children will be randomly and equally allocated into three groups, by throwing a dice (1&4 for group A, 2&5 for group B and 3&6 for group C). 10 for each group as follows: -

* Group A (Isobutyl cyanoacrylate): 10 children will be treated with isobutyl cyanoacrylate high viscous solution will be applied on the ulcer site.
* Group B (control positive): 10 children will be treated with chlorhexidine (0.2%) gel twice daily for 9 days.
* Group C (control negative): 10 children will be treated with normal saline will be applied on the ulcer site 5 times per day.

  * Children will be examined before treatment to assess pain by using Children's International Mucositis Evaluation Scale (ChIMES) and measure ulcer size by periodontal probe. Then apply different treatments of each group
  * All patients in both groups will be instructed to avoid eating or drinking for at least half an hour after oral administration of the oral gel.
  * All patients can be given oral analgesics (paracetamol) if needed to decrease pain severity.
  * The size of the ulcers, change in pain severity will be assessed on the 1st, 5th and 9th days after using isobutyl cyanoacrylate high viscous solution and chlorhexidine (0.2%) gel.

Assessment of pain will be performed using Children's International Mucositis Evaluation Scale (ChIMES) will be used for pain assessment

1. Photographs of the ulcers will be recorded with a digital camera at 1st, 5th and 9th days.
2. Measurement of ulcer size by using a periodontal probe

ELIGIBILITY:
Inclusion Criteria:

Apparently healthy cooperative children free from any systemic diseases that may predispose oral ulceration.

Development of pain/ulceration in the oral mucosa, surrounded by light red areola less than 1 cm. diameter.

Child with good oral hygiene. Parents willing to participate in the study and have a good likelihood of recall availability

Exclusion Criteria:

Taking of drugs that may influence the pattern of oral ulceration Oral ulcerations with unknown etiology that are not traumatic in nature. Allergic or who have suffered adverse reactions to isobutyl cyanoacrylate gel or chlorhexidine gel

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2024-08-04 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
pain assessment | 1st, 5th and 9th days
  Assessment of pain will be performed using Children's International Mucositis Evaluation Scale (ChIMES)
Measurement of ulcer size | 1st, 5th and 9th days.
  Photographs of the ulcers will be recorded with a digital camera and Measurement of ulcer size by using a periodontal probe.

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No